CLINICAL TRIAL: NCT01212393
Title: Prevention of Venous Thromboembolism Disease for Acutelly Ill Medical Patients Admitted to Hospital : Systematic Analysis of Thrombosis Risk Factors and Remember of Prevention Treatment Indications in Emergency Departments.
Brief Title: Prevention of Venous Thromboembolism Disease in Emergency Departments
Acronym: PREVENU
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHRC 2008-02
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2016-12

CONDITIONS: Quality of Health Care
Keywords: venous thromboembolism disease; emergency; prevention; thromboprophylaxis; medical; hosptitalization; health care risks
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — observational study at the patient level - cluster randomized study
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Intervention group: reminders
  Interventions: Behavioral: reminders
- current practice group: no intervention

INTERVENTIONS:
Behavioral: reminders — In the intervention group, emergency departments will be provided with poster and pocket cards and, if possible, with a computer decision support system remembering venous thromboembolism prophylactic treatment.
  Groups: Intervention group

SUMMARY:
The appropriate use of thromboprophylaxis in medical patients admitted to hospital can substantially reduce the overall burden of disease due to venous thromboembolism. However, the use of thromboprophylaxis in medical setting appears to be generally poor leaving at-risk patients unprotected.

We aim to analyse the incidence of symptomatic thromboembolic disease following hospitalisation in medical setting and the efficacy of a multicomponent prevention approach in emergency department including systematic evaluation of thrombosis risk factors and remembers of thrombophylaxis indications and modalities for acutely ill medical patients.

Design: cluster randomized interventional study - Observational study at patient level

Setting: 30 French emergency departments

Patients: Patients over 40 years old admitted in participating emergency departments and hospitalized for acute medical reasons.

Main judgment criteria: the rate of symptomatic thromboembolic events and severe haemorrhage during a formal 3-months follow-up after hospital admission in patients hospitalized at least 48 hours.

DETAILED DESCRIPTION:
Method:

At the end of an observational period of a week, centers will be randomized in two groups: intervention or current practice. In the intervention group, centers will be provided with poster and pocket cards and, if possible, with a computer decision support system remembering venous thromboembolism prophylactic treatment. We will propose no change in current practice in the other group.

Primary outcome: the rate of symptomatic venous thromboembolic events and severe haemorrhage during a formal 3-months follow-up after hospital admission in patients hospitalized at least 48 hours.

All possible thromboembolic events, severe haemorrhages and deaths will be analysed by an adjudication committee blinded of group assignation. Sudden death without obvious cause according to the adjudication committee will be considered as possible fatal pulmonary embolism.

Sample size: We calculated sample size on the basis of primary outcome. Assuming the participation of 30 centers (15 in each group), an intracluster correlation of 0.01, a rate of symptomatic thromboembolic events or severe haemorrhage of 5% in the current practice group, we need a sample of 16170 patients (8085 in each group) to detect a 1.5 percentage absolute difference between the 2 groups (3.5% in the intervention group) with a power of 80% and a significance level of 5%.

Considering a rate of patients hospitalized less than 48 hours around 5% and of lost of follow-up around 3%, we anticipated to include 16500 patients for the main analysis and 18000 patients for the overall study.

Secondary outcomes:

* The appropriateness of thromboprophylaxis in the overall population and according to group assignation:

  * Number of patients needing prevention treatment according to international recommendations and who have an appropriate treatment.
  * Number of patients without indication of thromboprophylaxis and who do not receive a treatment
* The rate of symptomatic venous thromboembolic events during a formal 3-months follow-up after hospital admission

  * in all included patients
  * in patients hospitalized at least 48 hours.
  * inpatients hospitalized less than 48 hours
* The rate of thromboembolic events

  * in patients who had an appropriate thromboprophylactic treatment
  * in patients who had an inappropriate thromboprophylactic treatment
  * in patients who had no thromboprophylactic treatment
* The rate of severe haemorrhage

  * in patients who had an appropriate thromboprophylactic treatment
  * in patients who had an inappropriate thromboprophylactic treatment
  * in patients who had no thromboprophylactic treatment

ELIGIBILITY:
Inclusion Criteria:

* age over 40 years
* Emergency department admission for non-traumatic reason
* Hospitalization in medical setting

Exclusion Criteria:

* patients less than 40 years old
* patients hospitalized in a facility which doesn't participate to the study
* 3 months follow-up not possible
* patients refusing that their personal data are used for medical research
* patients refusing to be reach for the 3 months follow-up

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible centers: Emergency departments previously implicated in research on venous thromboembolism.
  Eligible patients: patients over 40 years old admitted in participating emergency departments for non traumatic reason
Sampling Method: Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Symptomatic venous thromboembolic events and severe haemorrhage | 3 months
  the rate of symptomatic venous thromboembolic events and severe haemorrhage during a formal 3-months follow-up after hospital admission in patients hospitalized at least 48 hours.
  All possible thromboembolic events, severe haemorrhages and deaths will be analysed by an adjudication committee blinded of group assignation. Sudden death without obvious cause according to the adjudication committee will be considered as possible fatal pulmonary embolism.

SECONDARY OUTCOMES:
Rate of symptomatic venous thromboembolic events | 3 months
  - The rate of symptomatic venous thromboembolic events during a formal 3-months follow-up after hospital admission oin all included patients oin patients hospitalized at least 48 hours. oin patients hospitalized less than 48 hours
Rate of thromboembolic events | 3 months
  - The rate of thromboembolic events oin patients who had an appropriate thromboprophylactic treatment oin patients who had an inappropriate thromboprophylactic treatment oin patients who had no thromboprophylactic treatment
rate of severe haemorrhage | 3 months
  - The rate of severe haemorrhage oin patients who had an appropriate thromboprophylactic treatment oin patients who had an inappropriate thromboprophylactic treatment oin patients who had no thromboprophylactic treatment
appropriateness of thromboprophylaxis | 3 months
  - The appropriateness of thromboprophylaxis in the overall population and according to group assignation:
  oNumber of patients needing prevention treatment according to international recommendations and who have an appropriate treatment.
  oNumber of patients without indication of thromboprophylaxis and who do not receive a treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Marie ROY, MD, PhD, Principal Investigator — UH Angers
Locations (23):
- France (23):
  - UH Agen, Agen
  - H Argenteuil, Argenteuil
  - UH Besançon, Besançon
  - H Bethune, Béthune
  - H Bobigny, Bobigny
  - UH Ambroise Pare, Boulogne-Billancourt
  - UH Brest, Brest
  - H Chateauroux, Châteauroux
  - H Clermont Ferrand, Clermont-Ferrand
  - H Compiegne, Compiègne
  - UH Dijon, Dijon
  - UH Grenoble, Grenoble
  - UH La Reunion, La Réunion
  - UH Marseille, Marseille
  - UH Metz Thionville, Metz
  - UH Nantes, Nantes
  - UH Nimes, Nîmes
  - UH la pitié salpetriere, Paris
  - H Cochin, Paris
  - UH Bichat, Paris
  - UH Hotel Dieu, Paris
  - UH Poitiers, Poitiers
  - UH Rennes, Rennes

REFERENCES:
- [Derived] Roy PM, Rachas A, Meyer G, Le Gal G, Durieux P, El Kouri D, Honnart D, Schmidt J, Legall C, Hausfater P, Chretien JM, Mottier D; PREVENU study group. Multifaceted Intervention to Prevent Venous Thromboembolism in Patients Hospitalized for Acute Medical Illness: A Multicenter Cluster-Randomized Trial. PLoS One. 2016 May 26;11(5):e0154832. doi: 10.1371/journal.pone.0154832. eCollection 2016. PMID 27227406